CLINICAL TRIAL: NCT02381431
Title: Use of Mobile Phones for Thermal Imaging of the Chest to Save Lives of Children With Pneumonia in Nagpur, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Global Health, MGHfC, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P000265
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Infections - Bacterial; Pneumonia - Bacterial
Keywords: imaging; diagnostic; pediatrics
MeSH Terms: conditions — Bacterial Infections; Pneumonia, Bacterial; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermal Imaging (Experimental): imaging using a thermal camera
  Interventions: Device: FLIR ONE

INTERVENTIONS:
Device: FLIR ONE

SUMMARY:
The purpose of this study is to see if thermal images can be used instead of a chest x-ray to diagnose bacterial pneumonia in children with signs and symptoms of pneumonia in Nagpur, India. More specifically, the objectives of the study are: 1) to determine if thermal imaging, using a commercial thermal camera can accurately detect the presence of bacterial pneumonia in children receiving a chest x-ray to rule out pneumonia; 2) to evaluate the use of thermal imaging to monitor the course and resolution of pneumonia in children diagnosed with pneumonia; and 3) to determine if thermal imaging can accurately diagnose sites of infection that are suspected to be related to the pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or younger
* patient at DAGA Memorial Hospital, Nagpur, India
* had chest x-ray within last 24 hours
* consent obtained from one parent
* assent obtained if child is 8 years or older

Exclusion Criteria:

* thermal image cannot be done within 24 hours of chest x-ray

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
diagnosis of bacterial pneumonia | 24 hours
  Thermal imaging will be used and compared to the chest x-ray taken within 24 hours to see if bacterial pneumonia is present

SECONDARY OUTCOMES:
diagnosis of additional site of infection possibly related to bacterial pneumonia | within same hospital stay
  Thermal imaging will be used to image other potential sites of infection suspected of being related to the bacterial pneumonia if suspected by physician

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- DAGA Memorial Hospital, Nagpur, Maharashtra, India